CLINICAL TRIAL: NCT06319664
Title: Clinical Outcomes and Decision-making Choice of Skull Base Approaches for Petroclival Meningiomas: a Single Center Report of 179 Cases
Brief Title: Clinical Outcomes and Decision-making Choice of Skull Base Approaches for Petroclival Meningiomas
Status: Completed | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: sjnkzzj
Record Dates: First submitted 2024-01-17; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2021-03

CONDITIONS: Skull Base Meningioma
Keywords: clinical outcomes; petroclival meningioma; skull base approach; meningioma classification; operative technique

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Clivus type: The dural attachment originates from petroclival fissure, and the main portion of lesion is situated on middle-upper clivus, mainly grows toward the median line and even the heterolateral direction, could involve in the whole clivus region from dorsum sellae to foramen magnum.
  Interventions: Procedure: retrosigmoid approach (RSA)
- Petroclival type: The dural attachment originates likewise from petroclival fissure, but primarily extends toward the homolateral dorsal petrosum region, and the main portion is center on middle-upper clivus and grows toward petrous apex region forward and cerebellopontine angle region backward, leading to the homolateral trigeminus being compressed outwards.
  Interventions: Procedure: retrosigmoid approach (RSA)
- Petroclivosphenoidal type: The site of origin lies on petroclival region, while the main part of lesion is located in posterior cranial fossa and extends forward and upward along petroclival fissure, and could spread to posterior clinoid process, dorsum sellae and parasellar area with striding petrous ridge, or expanding into Meckel's cave (MC) and even reaching posterior wall of cavernous sinus (CS) through MC. Overall, the growth pattern direction is basically from posterior cranial fossa to middle cranial fossa and from the infratentorial to supratentorial compartment.
  Interventions: Procedure: retrosigmoid approach (RSA); Procedure: subtemporal transtentorial transpetrosal approach (STTA)
- Sphenopetroclival Subtype I: Sphenopetroclival type (S-PC type): The site of origin saddles the petrous ridge and invades the CS and parasellar region widely. The growth pattern is different from the PC-S type, mainly from the middle cranial fossa to the posterior cranial fossa. This type is then further classified into two subtypes based on the relationship between CS and the lesion site of origin. Subtype I (S-PC I type): The lesion mainly originates from posterior part of CS and posterior clinoid process region, could invade and break though the CS wall, and the main part of lesion expands towards parasellar, middle cranial fossa, and petrous apex, even invades the dorsum sellae and posterior cranial fossa through tentorium. As a result, the CS wall is mostly rough, and the dural space between the lesion and the temporal lobe is not well-defined on MRI.
  Interventions: Procedure: extended pterional transtentorial approach (EPTA); Procedure: presigmoid combined supra-infratentorial approach (PCA)
- Sphenopetroclival Subtype II: The dural attachment of lesion entirely originates within the CS leading to CS region expansile hyperplasia with the virtually intact sinus wall, and part of lesion could spread into the petrous apex and posterior cranial fossa through posterior sinus wall; the large partial lesions may also encroach on the lateral wall of the CS expansion towards the middle cranial fossa. The lateral sinus wall is relatively smooth and maintains the dural space between the lesion and the temporal lobe on MRI.
  Interventions: Procedure: pretemporal trancavernous anterior transpetrosal approach (PTCA); Procedure: presigmoid combined supra-infratentorial approach (PCA)
- Central Skull Base type: The dural attachment originates from the petroclival fissure, but growth pattern is widespread invasion of central skull base region and structures bilaterally and the site of origin extensively involves in dorsum sellae, clivus and bilateral suprasellar, parasellar and CS areas even cerebellopontine angle region.
  Interventions: Procedure: inoperable

INTERVENTIONS:
Procedure: retrosigmoid approach (RSA) — The skull base approach choice was fundamentally followed by the modified classification.
  Groups: Clivus type; Petroclival type; Petroclivosphenoidal type
Procedure: subtemporal transtentorial transpetrosal approach (STTA) — The skull base approach choice was fundamentally followed by the modified classification.
  Groups: Petroclivosphenoidal type
Procedure: extended pterional transtentorial approach (EPTA) — The skull base approach choice was fundamentally followed by the modified classification.
  Groups: Sphenopetroclival Subtype I
Procedure: pretemporal trancavernous anterior transpetrosal approach (PTCA) — The skull base approach choice was fundamentally followed by the modified classification.
  Groups: Sphenopetroclival Subtype II
Procedure: presigmoid combined supra-infratentorial approach (PCA) — The skull base approach choice was fundamentally followed by the modified classification.
  Groups: Sphenopetroclival Subtype I; Sphenopetroclival Subtype II
Procedure: inoperable — The skull base approach choice was fundamentally followed by the modified classification.
  Groups: Central Skull Base type

SUMMARY:
Petroclival meningioma (PCM) is a technically challenging lesion. We aimed to analyze the role of various skull base approaches and evaluate the therapeutic outcomes guided by the modified classification. We retrospectively analyzed the clinical characteristics, surgical approaches, outcomes and follow-up data from 179 cases of PCM from January 2011 to December 2020. We modified the previous classification into updated five types with two subtypes: clivus type (CV), petroclival type (PC), petroclivosphenoidal type (PC-S), sphenopetroclival type (S-PC) with two subtypes of S-PC I and S-PC II and central skull base type (CSB). Statistical analysis was performed using IBM SPSS Statistical Package 21.0. The t-test was performed to clinical data comparisons between the two groups and the ANOVA test was used to compare the difference between multiple groups. P < 0.05 was considered statistically significant.

DETAILED DESCRIPTION:
1. Study Design and Ethics Approval In this institutional study, 179 cases of PCM were retrospectively collected and analyzed from January 2011 to December 2020 in our neurosurgical department, Xiangya Hospital, Central South University. The studies involving human participants were reviewed and approved by the Ethics Committee of Xiangya Hospital, Central South University (approval no. 202103227) in accordance with the ethical standards of the 1964 Declaration of Helsinki and its later amendments. Patients provided their written informed consent to participate in this study. Written informed consent was obtained from the individual(s) for the publication of any potentially identiﬁable images or data included in this article.
2. Evaluative Criteria Clinical characteristics with manifestation, neurological function status, neuroimaging and surgical records, and follow-up data were reviewed and evaluated. The preoperative, postoperative and follow-up QOL were assessed and measured using the Karnofsky Performance Scale (KPS) score by two neurosurgeons, independently, on admission, discharge, and follow-up, correspondingly. The preoperative radiological data were obtained from routine examination of brain 3.0 T magnetic resonance imaging (MRI) with T1-weighted, T2-weighted and T1-contrast-enhanced sequences, computed tomography angiography (CTA) and skull base high-resolution computed tomography (HRCT) scans to evaluate tumor size, origin of dural attachment, growth pattern, involved circumjacent range, brainstem displacement, peritumoral edema, encasement of vital neurovascular structure and hydrocephalus to further identify tumor classification and treatment strategy. All of cases were re-examined with contrast MRI to identify the EOR within 72 hours post-operative. The EOR was divided into three levels of gross total resection (GTR) (Simpson Grades I/II), subtotal resection (STR) (Simpson Grades III/IV, with 90-99% excision of the lesion) and partial resection (PR) (Simpson III/IV, with below 90% excision of the lesion), depending on the intraoperative identification and postoperative MRI.

   A combination of outpatient, telephone and Internet connections were used for follow-up. Follow-up data, including clinical and radiographic information, was collected 3 and 6 months after the surgical procedure and then every 1 or 2 years, in most cases via clinic visits. Questionnaires and phone calls were also carried out. The tumor recurrence or progress (R/P) meant lesion regrowth in situ in GTR cases or residual lesion regrowth with the increase of the maximal diameter more than 3 mm in STR/PR cases. Those who experienced tumor R/P were recommended for additional treatment. The latest follow-up deadline is March 1, 2021.
3. PCM Classification On the basis of the variation of PCM pathological alteration in anatomy and with the accumulating experience and incisive comprehension to PCM, we modified and improved our previous tumor classification into updated five types with two subtypes: clivus type (CV), petroclival type (PC), petroclivosphenoidal type (PC-S), sphenopetroclival type (S-PC) with two subtypes of S-PC I and S-PC II and central skull base type (CSB).
4. Skull Base Approach Choice The skull base approach choice was fundamentally followed by the modified classification. At the same time, the patient's age, request and physical condition cannot be ignored. In this study, the retrosigmoid approach (RSA), subtemporal transtentorial transpetrosal approach (STTA), extended pterional transtentorial approach (EPTA), pretemporal trancavernous anterior transpetrosal approach (PTCA) and presigmoid combined supra-infratentorial approach (PCA) were applied as the main surgical approaches. Moreover, the RSA included basic retrosigmoid approach (BRSA), retrosigmoid trantentorial approach (RTTA) and retrosigmoid intradural suprameatal approach (RISA). Intraoperative neurophysiological monitoring containing somatosensory evoked potentials (SSEP), motor evoked potentials (MEP) and brainstem auditory evoked potentials (BAEP) were essentially and routinely implemented.
5. Statistical Analysis Statistical analysis was performed using IBM SPSS Statistical Package 21.0. The t-test was performed to clinical data comparisons between the two groups and the ANOVA test was used to compare the difference between multiple groups. P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as the PCM from the MRI follwoed the definition of PCM.

Exclusion Criteria:

* 1. combined with serious chronic diseases leading to inoperable therapy; 2. the partient refused to recevie surgical therapy; 3. combined with other cancers.

Ages: 15 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In this institutional study, 179 cases of PCM were retrospectively collected and analyzed from January 2011 to December 2020 in our neurosurgical department, Xiangya Hospital, Central South University. This study enrolled 28 males and 151 females with a male to female ratio of 1:5.4 and average age of 49.9±10.2 years (range 15-73 years). A total of 16 cases (8.9%) had been treated in other hospitals preoperatively with 12 cases of prior operations and 4 cases of prior gamma knife radiosurgery (GKS).
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
QOL were assessed and measured using the Karnofsky Performance Scale (KPS) score | an average of 1 year
  QOL were assessed and measured using the Karnofsky Performance Scale (KPS) score by two neurosurgeons, independently, on admission, discharge, and follow-up, correspondingly. Follow-up KPS score was collected through study completion, an average of 1 year, in most cases via clinic visits.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Liu, MD, Study Director — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
When the research data has been published.

REFERENCES:
- [Result] Research must do no harm: new guidance addresses all studies relating to people. Nature. 2022 Jun;606(7914):434. doi: 10.1038/d41586-022-01607-0. No abstract available. PMID 35701624